CLINICAL TRIAL: NCT03296904
Title: The CYBERnetic LowEr-Limb CoGnitive Ortho-prosthesis Plus Plus, 1st Clinical Study: Validation of the Efficacy of the CYBERnetic LowEr-Limb CoGnitive Ortho-prosthesis Plus Plus Modules in a Clinical Setting
Brief Title: The CYBERnetic LowEr-Limb CoGnitive Ortho-prosthesis Plus Plus, 1st Clinical Study
Acronym: CLs++1stCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other); Université Catholique de Louvain (Other); Vrije Universiteit Brussel (Other); University of Ljubljana (Other); Össur Iceland ehf (Industry); IUVO Srl (Unknown)
Responsible Party: Principal Investigator, Raffaele Molino Lova, MD, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYBERLEGs Plus Plus
Record Dates: First submitted 2017-09-19; First posted 2017-09-29 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Transfemoral Amputation
Keywords: Lower limb amputation; Wearable robotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLs++ (Experimental): Baseline assessment, intervention, final assessment
  Interventions: Device: CLs++

INTERVENTIONS:
Device: CLs++ — Familiarization/training with the customized combination of the CLs++ ortho-prosthesis modules

SUMMARY:
The global goal of the CYBERnetic LowEr-limb coGnitive ortho-prosthesis Plus Plus (CLs++) project is to validate the technical and economic viability of the powered robotic ortho-prosthesis developed within the 7th Framework Program - Information and Communication Technology - CYBERnetic LowEr-limb coGnitive ortho-prosthesis project, as a means to enhance/ restore the mobility of transfemoral amputees and to enable them to perform locomotion tasks such as ground-level walking, climbing/descending stairs, standing up, sitting down and turning in scenarios of real life. Restored mobility will allow amputees to perform physical activity thus counteracting physical and cognitive decline which occurs with advancing age and improving the overall health status and quality of life.

This project involves players from academia, research institutions, end users, as well as robotics and healthcare industry, and has been funded by the European Commission (call identifier H2020 - Information and Communication Technology 24-2015, scope c, namely Technology Transfer - Robotics use cases, Grant Agreement 731931).

The CLs++ project is an Innovation Action (IA) and foresees 2 clinical studies aimed at assessing the efficacy of the CLs++ modules in different settings.

In this 1st clinical study, 16 patients with unilateral trans-femoral amputation, 8 @ the Don Gnocchi Foundation, Center of Florence, and 8 @ the Free University of Brussels, Dept. of Human Physiology, will participate in the assessment of the efficacy of the CLs++ ortho-prosthesis modules in a clinical setting.

DETAILED DESCRIPTION:
In the first clinical study, a set of combinations of the three hardware (HW) modules of the CLs++ ortho-prosthesis, namely the Active Trans-femoral Prosthesis (ATP), the Active Pelvis Orthosis (APO) and the Active Knee Orthosis (AKO) will be tested, along with the Wearable Sensory Apparatus (WSA), the Bidirectional Interface (BI) and the control software (SW).

The recruitment of potential participants will be carried out by a multidisciplinary team (physicians, physiotherapists and psychologists) and will be aimed at ascertaining the inclusion and exclusion criteria as reported in the "Eligibility" section. If the potential participant fulfills the requirements to be enrolled, the responsible for the study will provide him/her with the information sheet and will answer all possible questions. Once the participant agrees to participate in the study, he/she will sign the informed consent form. An appointment will also be arranged with the orthopedic workshop to make a spare socket to be used with the ATP.

The protocol of the CLs++ first clinical study will be constituted by two main phases.

The first phase is expected to last one week and it has the goal to explore the functionality of the CLs++ HW and SW modules in structured or semi-structured clinical settings by means of a preliminary initial set of activities. In particular, the enrolled participants will be testing 4 different combinations of CLs++ modules:

a) APO + WSA + BI; b) ATP + WSA; c) APO + ATP + WSA; d) APO + AKO + WSA.

This set of experiments will allow to collect relevant data at the beginning of the protocol in order to assess the functionality of the CLs++ system for each participant. Furthermore, the appropriate combination of the three HW modules of the CLs++ ortho-prosthesis will be selected among one of the above combinations. The selection will be performed with participants walking overground and on a treadmill at their self-selected speed, to optimally match the specific user needs based on their residual movement ability and required movement assistance. Specifically, the appropriate combination of the CLs++ modules will be selected based on both the clinical evaluation (e.g. walking asymmetry, stump length, flexion-extension hip strength, strength of the contra-lateral limb) and the subjective feedback, in terms of comfort and perceived functionality, from the participant.

Assessments will be performed at the beginning and at the end of the 1-month familiarization/training period, with participants wearing both their customized combination of the CLs++ modules and their own prosthesis only. The functional assessments will be performed using a treadmill to be able to control all variables: however, we will also perform some test during over-ground walking. In addition to the assessments reported in the section "Outcome Measures", the study foresees the administration of the System Usability Scale (SUS) to assess the usability of the CLs++ system. The study also foresees the development of ad-hoc tools for investigating the economic dimension.

The second phase of the study will consist of an hospital-based familiarization/training walking on the treadmill and overground with the selected combination of CLs++ modules, 1 hour 3 times a week for 1 month. Worthily, training sessions will be mainly focused on the familiarization to the use of the customized combination of CLs++ modules rather than on aerobic training. Thus, the work load, as expressed by the walking speed overground or on the treadmill, will not be critical. Further, participants will be asked to walk at their self-selected speed and will be allowed to stop walking whenever they feel tired and to start again walking once they have recovered.

After 2 weeks of familiarization/training, the set of assessments can be repeated in order to assess whether the experience gained in the training period has effects on a different set of CLs++ modules. Notably, the initial set of modules identified for each patient will be kept unchanged for the whole duration of the familiarization/training, and the intermediate session will be used as evaluation means.

From a statistical point of view, as reported in the "Study Design" section, a sample size of 16 subjects will be able to detect a 15% change in walking-related physical effort, in terms of oxygen uptake during the six-minute walk test, in a single group of trans-femoral amputees with a statistical power > 0.9 at the two-sided 0.05 alpha-level. Descriptive statistics will be used to present results, while appropriate inferential statistics will be used to ascertain possible significant differences. Data will be also analysed following a case-series approach: data of each patient will be analysed separately in order to highlight the occurrence of differences between pre- and post- assessment sessions, or any learning effect over the familiarization/training time.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral trans-femoral amputation (any cause)
* Completed the post amputation rehabilitation process
* Medicare Functional Classification Level ≤ K3

Exclusion Criteria:

* Poor cognitive skills (Mini Mental State Examination)
* Severe anxiety or depression (State-Trait Anxiety Inventory Form Y and Beck Depression Inventory II, respectively)
* Relevant comorbidity (hemiplegia, degenerative nervous system diseases, hip or knee replacement, chronic heart failure, chronic obstructive pulmonary disease, act.)
* Stump pain/socket poor fitting
* Implantable cardiac devices (PMK and AICD)
* Inability to walk on a treadmill

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in the physical effort needed for walking with the participant's own prosthesis vs. with the customized combination of CLs++ ortho-prosthesis modules. | Before and after the familiarization/training period lasting one month.
  While performing the six-minute walk test, oxygen uptake will be assessed using a portable gas analyzer and will be considered as an objective measure of the physical effort.

SECONDARY OUTCOMES:
Change in the self-perceived physical effort needed for walking with the participant's own prosthesis vs. with the customized combination of CLs++ ortho-prosthesis modules. | Before and after the familiarization/training period lasting one month.
  At the end of the six-minute walk test, the Borg Scale (CR-10) will be administered and the score will be considered as a measure of the perceived physical effort.
Change in the cognitive effort needed for walking with the participant's own prosthesis vs. with the customized combination of CLs++ ortho-prosthesis modules | Before and after the familiarization/training period lasting one month.
  The cognitive effort will be assessed through changes in the galvanic skin response (GSR), heart rate variability (HRV) and brain electrical activity (EEG) while performing two Dual Task tests, namely the backward counting and the Stroop test.
Change in the performance during stair climbing/descending with the participant's own prosthesis vs. with the customized combination of CLs++ ortho-prosthesis modules. | Before and after the familiarization/training period lasting one month.
  The performance in the above locomotion-related task will be assessed using the Stair Climbing Test (SCT).
Change in the performance during sitting down/standing-up and turning with the participant's own prosthesis vs. with the customized combination of CLs++ ortho-prosthesis modules | Before and after the familiarization/training period lasting one month.
  The performance in the above locomotion-related task will be assessed using the Timed get-Up and Go test (TUG)
Change in gait asymmetry with the participant's own prosthesis vs. with the customized combination of CLs++ ortho-prosthesis modules | Before and after the familiarization/training period lasting one month.
  Gait asymmetry will be assessed using a motion capture system, either optoelectronic or marker-less.
Change in muscle electrical activity with the participant's own prosthesis vs. with the customized combination of CLs++ ortho-prosthesis modules | Before and after the familiarization/training period lasting one month.
  Muscle electrical activity will be assessed using surface electromyography (sEMG)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Molino Lova, MD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi Onlus, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monaco V, Tropea P, Aprigliano F, Martelli D, Parri A, Cortese M, Molino-Lova R, Vitiello N, Micera S. An ecologically-controlled exoskeleton can improve balance recovery after slippage. Sci Rep. 2017 May 11;7:46721. doi: 10.1038/srep46721. PMID 28492520
- [Background] d'Elia N, Vanetti F, Cempini M, Pasquini G, Parri A, Rabuffetti M, Ferrarin M, Lova RM, Vitiello N. Erratum to: Physical human-robot interaction of an active pelvis orthosis: toward ergonomic assessment of wearable robots. J Neuroeng Rehabil. 2017 Jun 5;14(1):51. doi: 10.1186/s12984-017-0262-x. No abstract available. PMID 28583163
- [Background] Ruiz Garate V, Parri A, Yan T, Munih M, Molino Lova R, Vitiello N, Ronsse R. Experimental Validation of Motor Primitive-Based Control for Leg Exoskeletons during Continuous Multi-Locomotion Tasks. Front Neurorobot. 2017 Mar 17;11:15. doi: 10.3389/fnbot.2017.00015. eCollection 2017. PMID 28367121
- [Background] Zheng E, Manca S, Yan T, Parri A, Vitiello N, Wang Q. Gait Phase Estimation Based on Noncontact Capacitive Sensing and Adaptive Oscillators. IEEE Trans Biomed Eng. 2017 Oct;64(10):2419-2430. doi: 10.1109/TBME.2017.2672720. Epub 2017 Feb 23. PMID 28252387
- [Background] Motor primitive-based control for lower-limb exoskeletons Virginia Ruiz Garate, Andrea Parri , Tingfang Yan, Marko Munih, Raffaele Molino Lova, Nicola Vitiello, and Renaud Ronsse 6th IEEE RAS/EMBS International Conference on Biomedical Robotics and Biomechatronics (BioRob) June 26-29, 2016. U Town, Singapore, pag. 655-661.
- [Background] Walking Assistance using Motor Primitives Virginia Ruiz Garate, Andrea Parri, Tingfang Yan, Marko Munih, Raffaele Molino Lova, Nicola Vitiello, and Renaud Ronsse. IEEE Robotics and Automation Magazine 2014, March 2016, pag.83-95.
- [Background] Yuan K, Parri A, Yan T, Wang L, Munih M, Vitiello N, Wang Q. Fuzzy-logic-based hybrid locomotion mode classification for an active pelvis orthosis: Preliminary results. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:3893-6. doi: 10.1109/EMBC.2015.7319244. PMID 26737144
- [Background] Grazi L, Crea S, Parri A, Yan T, Cortese M, Giovacchini F, Cempini M, Pasquini G, Micera S, Vitiello N. Gastrocnemius myoelectric control of a robotic hip exoskeleton. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:3881-4. doi: 10.1109/EMBC.2015.7319241. PMID 26737141
- [Background] CYBERLEGs - A User-Oriented Robotic Transfemoral Prosthesis with Whole Body Awareness Control. Ambrožič L, Goršič M, Geeroms J, Flynn L, Molino Lova R, Kamnik R, Munih M, Vitiello N. IEEE Robotics and Automation Magazine 2014, vol. 21(4):82-93.
- [Background] Gorsic M, Kamnik R, Ambrozic L, Vitiello N, Lefeber D, Pasquini G, Munih M. Online phase detection using wearable sensors for walking with a robotic prosthesis. Sensors (Basel). 2014 Feb 11;14(2):2776-94. doi: 10.3390/s140202776. PMID 24521944
- See also: Official website of the CYBERnetic LowEr-limb coGnitive ortho-prosthesis Plus Plus project — http://www.cyberlegs.eu